CLINICAL TRIAL: NCT01133093
Title: Study on Nutrition and Cardiovascular Risk in Spain.
Acronym: ENRICA
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jose R Banegas, Professor of Preventive Medicine and Public Health, Universidad Autonoma de Madrid
Other Study IDs: ENRICA
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular risk factors; Nutritional assessment; Epidemiology
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the distribution, awareness and control of main cardiovascular risk factors in the Spanish population. The main study variables are:

* Lifestyles (tobacco, alcohol, nutrition, physical activity)
* Biological risk factors either well-established (blood lipids, glucose, insulin and blood pressure) or emergent (leptin, C-reactive protein and other markers of inflammation)

DETAILED DESCRIPTION:
Data collection comprised 3 sequential stages:

1. computer-assisted telephone interview to obtain information on lifestyle, knowledge and attitudes about cardiovascular disease risk factors, and the signs and symptoms of heart attack and stroke, subjective health, and morbidity;
2. first homevisit, to collect blood and urine samples for analysis by a central laboratory;
3. second home visit, to measure anthropometric variables and blood pressure and to administer a computer-assisted dietary history; data on functional limitations are also collected from participants aged 65 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized Spanish resident
* 18 years and over

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample representative of the non-institutionalized Spanish population
Sampling Method: Probability Sample
Enrollment: 11991 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk Factors Control | 2 years
Health-related quality of life | 2 years
Use of health care services | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Banegas, MD, PhD, Principal Investigator — Department of Preventive Medicine and Public Health, Universidad Autonoma de Madrid; Fernando Rodriguez-Artalejo, MD, PhD, Principal Investigator — Department of Preventive Medicine and Public Health, Universidad Autonoma de Madrid
Locations (1):
- Department of Preventive Medicine and Public Health. Universidad Autonoma de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gutierrez-Fisac JL, Guallar-Castillon P, Leon-Munoz LM, Graciani A, Banegas JR, Rodriguez-Artalejo F. Prevalence of general and abdominal obesity in the adult population of Spain, 2008-2010: the ENRICA study. Obes Rev. 2012 Apr;13(4):388-92. doi: 10.1111/j.1467-789X.2011.00964.x. Epub 2011 Dec 12. PMID 22151906
- [Result] Guallar-Castillon P, Gil-Montero M, Leon-Munoz LM, Graciani A, Bayan-Bravo A, Taboada JM, Banegas JR, Rodriguez-Artalejo F. Magnitude and management of hypercholesterolemia in the adult population of Spain, 2008-2010: The ENRICA Study. Rev Esp Cardiol (Engl Ed). 2012 Jun;65(6):551-8. doi: 10.1016/j.recesp.2012.02.005. Epub 2012 Apr 5. PMID 22483404
- [Result] Leon-Munoz LM, Guallar-Castillon P, Graciani A, Lopez-Garcia E, Mesas AE, Aguilera MT, Banegas JR, Rodriguez-Artalejo F. Adherence to the Mediterranean diet pattern has declined in Spanish adults. J Nutr. 2012 Oct;142(10):1843-50. doi: 10.3945/jn.112.164616. Epub 2012 Aug 8. PMID 22875552
- [Result] Banegas JR, Graciani A, de la Cruz-Troca JJ, Leon-Munoz LM, Guallar-Castillon P, Coca A, Ruilope LM, Rodriguez-Artalejo F. Achievement of cardiometabolic goals in aware hypertensive patients in Spain: a nationwide population-based study. Hypertension. 2012 Oct;60(4):898-905. doi: 10.1161/HYPERTENSIONAHA.112.193078. Epub 2012 Sep 4. PMID 22949530
- [Result] Mesas AE, Leon-Munoz LM, Guallar-Castillon P, Graciani A, Gutierrez-Fisac JL, Lopez-Garcia E, Aguilera MT, Banegas JR, Rodriguez-Artalejo F. Obesity-related eating behaviours in the adult population of Spain, 2008-2010. Obes Rev. 2012 Oct;13(10):858-67. doi: 10.1111/j.1467-789X.2012.01005.x. Epub 2012 May 11. PMID 22577840
- [Result] Lundelin K, Graciani A, Garcia-Puig J, Guallar-Castillon P, Taboada JM, Rodriguez-Artalejo F, Banegas JR. Knowledge of stroke warning symptoms and intended action in response to stroke in Spain: a nationwide population-based study. Cerebrovasc Dis. 2012;34(2):161-8. doi: 10.1159/000341408. Epub 2012 Aug 17. PMID 22907330
- [Result] Navarro-Vidal B, Banegas JR, Leon-Munoz LM, Rodriguez-Artalejo F, Graciani A. Achievement of cardiometabolic goals among diabetic patients in Spain. A nationwide population-based study. PLoS One. 2013 Apr 18;8(4):e61549. doi: 10.1371/journal.pone.0061549. Print 2013. PMID 23637851
- [Result] Graciani A, Leon-Munoz LM, Guallar-Castillon P, Rodriguez-Artalejo F, Banegas JR. Cardiovascular health in a southern Mediterranean European country: a nationwide population-based study. Circ Cardiovasc Qual Outcomes. 2013 Jan 1;6(1):90-8. doi: 10.1161/CIRCOUTCOMES.112.967893. Epub 2013 Jan 8. PMID 23300271
- [Result] Lopez-Garcia E, Guallar-Castillon P, Leon-Munoz L, Rodriguez-Artalejo F. Prevalence and determinants of metabolically healthy obesity in Spain. Atherosclerosis. 2013 Nov;231(1):152-7. doi: 10.1016/j.atherosclerosis.2013.09.003. Epub 2013 Sep 18. PMID 24125427
- [Result] Soler-Vila H, Galan I, Valencia-Martin JL, Leon-Munoz LM, Guallar-Castillon P, Rodriguez-Artalejo F. Binge drinking in Spain, 2008-2010. Alcohol Clin Exp Res. 2014 Mar;38(3):810-9. doi: 10.1111/acer.12275. Epub 2013 Oct 24. PMID 24164355
- [Result] Graciani A, Rodriguez-Artalejo F, Navarro-Vidal B, Banegas JR. Glycemic control using individualized targets among diabetic patients in Spain: a population-based study. Rev Esp Cardiol (Engl Ed). 2014 Feb;67(2):151-3. doi: 10.1016/j.rec.2013.07.018. Epub 2013 Dec 4. No abstract available. PMID 24795130
- [Result] Guallar-Castillon P, Perez RF, Lopez Garcia E, Leon-Munoz LM, Aguilera MT, Graciani A, Gutierrez-Fisac JL, Banegas JR, Rodriguez-Artalejo F. Magnitude and management of metabolic syndrome in Spain in 2008-2010: the ENRICA study. Rev Esp Cardiol (Engl Ed). 2014 May;67(5):367-73. doi: 10.1016/j.rec.2013.08.014. Epub 2014 Jan 14. PMID 24774729
- [Result] Leon-Munoz LM, Galan I, Donado-Campos J, Sanchez-Alonso F, Lopez-Garcia E, Valencia-Martin JL, Guallar-Castillon P, Rodriguez-Artalejo F. Patterns of alcohol consumption in the older population of Spain, 2008-2010. J Acad Nutr Diet. 2015 Feb;115(2):213-224. doi: 10.1016/j.jand.2014.08.017. Epub 2014 Oct 5. PMID 25288520
- [Derived] Blanco-Rojo R, Sandoval-Insausti H, Lopez-Garcia E, Graciani A, Ordovas JM, Banegas JR, Rodriguez-Artalejo F, Guallar-Castillon P. Consumption of Ultra-Processed Foods and Mortality: A National Prospective Cohort in Spain. Mayo Clin Proc. 2019 Nov;94(11):2178-2188. doi: 10.1016/j.mayocp.2019.03.035. Epub 2019 Oct 14. PMID 31623843
- [Derived] Laclaustra M, Rodriguez-Artalejo F, Guallar-Castillon P, Banegas JR, Graciani A, Garcia-Esquinas E, Lopez-Garcia E. The inflammatory potential of diet is related to incident frailty and slow walking in older adults. Clin Nutr. 2020 Jan;39(1):185-191. doi: 10.1016/j.clnu.2019.01.013. Epub 2019 Jan 24. PMID 30737049
- [Derived] Rodriguez-Artalejo F, Graciani A, Guallar-Castillon P, Leon-Munoz LM, Zuluaga MC, Lopez-Garcia E, Gutierrez-Fisac JL, Taboada JM, Aguilera MT, Regidor E, Villar-Alvarez F, Banegas JR. [Rationale and methods of the study on nutrition and cardiovascular risk in Spain (ENRICA)]. Rev Esp Cardiol. 2011 Oct;64(10):876-82. doi: 10.1016/j.recesp.2011.05.019. Epub 2011 Aug 6. Spanish. PMID 21821340